CLINICAL TRIAL: NCT00093912
Title: Evaluation of Clevidipine in the Perioperative Treatment of Hypertension Assessing Safety Events (With Sodium Nitroprusside as Active Comparator) (ECLISPE-SNP)
Brief Title: Clevidipine in the Perioperative Treatment of Hypertension (ECLISPE-SNP)
Acronym: ECLISPE-SNP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The Medicines Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TMC-CLV-03-04; ECLIPSE-SNP (Other: Sponsor)
Record Dates: First submitted 2004-10-07; First posted 2004-10-08 (Estimated); Last update posted 2014-05-06 (Estimated); Status verified 2014-05

CONDITIONS: Hypertension
Keywords: Perioperative Hypertension
MeSH Terms: conditions — Hypertension | interventions — clevidipine; Nitroprusside

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- clevidipine (Experimental): Clevidipine (0.5 mg/mL in 20% lipid emulsion) was initiated after insertion of an arterial line upon the occurrence of perioperative hypertension, as determined by the investigator, and was administered intravenously (IV) at an initial infusion rate of 0.4 μg/kg/min (non weight-based equivalent is 2 mg/h). Clevidipine was titrated to blood pressure lowering effect by doubling increments approximately every 90 seconds up to a maximum infusion rate of 3.2 μg/kg/min (16 mg/h). Infusion rates above 3.2 μg/kg/min were permitted up to the maximum infusion rate of 8.0 μg/kg/min. Treatment was maintained as long as was deemed clinically necessary or until discharge from the ICU. Infusion rates between 4.4 and 8.0 μg/kg/min were to be administered for no more than 2 hours.
  Interventions: Drug: clevidipine
- sodium nitroprusside (Active Comparator): Sodium nitroprusside (SNP) was initiated after insertion of an arterial line upon the occurrence of perioperative hypertension, as determined by the investigator, and was administered intravenously as per institutional practice. Treatment was maintained as long as was deemed clinically necessary or until discharge from the ICU.
  Interventions: Drug: sodium nitroprusside

INTERVENTIONS:
Drug: clevidipine
  Other Names: clevidipine, Cleviprex
  Arms: clevidipine
Drug: sodium nitroprusside
  Arms: sodium nitroprusside

SUMMARY:
The purpose of this study is to establish the safety of clevidipine in the treatment of perioperative hypertension. Approximately 250-500 patients with perioperative hypertension undergoing coronary artery bypass grafting (CABG), off-pump coronary artery bypass (OPCAB) or minimally invasive direct coronary artery bypass (MIDCAB) surgery and/or valve replacement/repair procedures were anticipated to be randomly assigned to one of two treatment groups: clevidipine or sodium nitroprusside.

DETAILED DESCRIPTION:
The primary objective was to establish the safety of clevidipine in the treatment of perioperative hypertension, as assessed by comparing the incidences of death, stroke, MI and renal dysfunction in the clevidipine and sodium nitroprusside treatment groups from the initiation of study drug infusion through postoperative Day 30. Secondary objectives were to evaluate the efficacy of study drug, assessed by the blood pressure (BP) lowering effect and additional safety variables.

ELIGIBILITY:
Prerandomization Inclusion Criteria:

* Provide written informed consent before initiation of any study related procedures.
* Be at least 18 years of age
* Be scheduled for Coronary Artery Bypass Grafting (CABG), Off Pump Coronary Artery Bypass (OPCAB), Minimally Invasive Direct Coronary Artery Bypass (MIDCAB) surgery, and/or valve replacement/repair surgery

Prerandomization Exclusion Criteria:

* Women of child-bearing potential (unless they have a negative pregnancy test)
* Recent cerebrovascular accident (within 3 months before randomization)
* Known intolerance to calcium channel blockers
* Known or suspected hypersensitivity to sodium nitroprusside
* Allergy to soybean oil or egg lecithin (components of the lipid vehicle)
* Pre-existing permanent ventricular pacing
* Any other disease or condition, which, in the judgment of the investigator would place a patient at undue risk by being enrolled in the trial
* Participation in another therapeutic drug or therapeutic device trial within 30 days of starting study

Postrandomization Inclusion Criteria:

* Determined to be hypertensive perioperatively as determined by the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 739 (Actual)
Dates: Start 2004-06; Primary Completion 2006-10 (Actual); Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Incidence of death, stroke, MI and renal dysfunction | Initiation of study drug infusion through post-operative Day 30

CONTACTS AND LOCATIONS:
Overall Officials: Malcolm Lloyd, MD, Study Director — The Medicines Company - Medical Director, Clinical Operations
Locations (29):
- United States (29):
  - Saint Vincents Hospital, Birmingham, Alabama
  - Brookwood Medical Center, Birmingham, Alabama
  - Baptist Medical Center, Montclair, Birmingham, Alabama
  - Baptist Medical Center, South, Montgomery, Alabama
  - Drug Research and Analysis Corporation, Montgomery, Alabama
  - Providence Saint Joseph Medical Center, Burbank, California
  - Stanford University Medical Center, Stanford, California
  - Shands Hospital at the University of Florida, Gainesville, Florida
  - Health First Holmes Regional Medical Center, Melbourne, Florida
  - Kaiser Permanente, Honolulu, Hawaii
  - St. Francis Hospital and Health Center, Blue Island, Illinois
  - St. Francis Hospital of Evanston, Evanston, Illinois
  - Wesley Medical Center, Wichita, Kansas
  - Touro Infirmary, New Orleans, Louisiana
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - St. Joseph Medical Center, Towson, Maryland
  - Massachussettes General Hospital, Boston, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - Saint Lukes Hospital, Duluth, Minnesota
  - International Heart Institute/St. Patrick Hospital, Missoula, Montana
  - Mt. Sinai Medical Center, New York, New York
  - The Christ Hospital, Cincinnati, Ohio
  - Portland VA Medical Center, Portland, Oregon
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Jackson-Madison County General Hospital, Jackson, Tennessee
  - Houston Northwest Medical Center, Houston, Texas
  - LDS Hospital, Salt Lake City, Utah
  - Virginia Commonwealth University Medical Center, Richmond, Virginia
  - Medical College of Wisconsin VAMC - Milwaukee, Milwaukee, Wisconsin

REFERENCES:
- [Result] Aronson S, Dyke CM, Stierer KA, Levy JH, Cheung AT, Lumb PD, Kereiakes DJ, Newman MF. The ECLIPSE trials: comparative studies of clevidipine to nitroglycerin, sodium nitroprusside, and nicardipine for acute hypertension treatment in cardiac surgery patients. Anesth Analg. 2008 Oct;107(4):1110-21. doi: 10.1213/ane.0b013e31818240db. PMID 18806012